CLINICAL TRIAL: NCT00437632
Title: A Placebo Controlled, Single Blind, Randomised Study Investigating the Safety, Tolerability and Pharmacokinetics of Repeated Oral Doses of GSK598809 in Healthy Male and Female Volunteers for 28 Days.
Brief Title: Study To Investigate If Repeat Doses Of GSK598809 Are Safe And Well Tolerated And To Evaluate Blood Levels Of GSK598809
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: DAN106587
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Substance Dependence
Keywords: repeat dose,; placebo,; Safety,; pharmacodynamics,; tolerability,; GSK598809; pharmacokinetics,
MeSH Terms: conditions — Substance-Related Disorders | interventions — GSK598809; Caffeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Subjects in Cohort-1 of Section 1 (Experimental): Subjects will be randomized to receive either GSK598809 10 mg or Placebo.
  Interventions: Drug: GSK598809; Drug: Placebo
- Subjects in Cohort-2 of Section 1 (Experimental): Subjects will be randomized to receive either GSK598809 25 mg or Placebo.
  Interventions: Drug: GSK598809; Drug: Placebo
- Subjects in Cohort-3 of Section 1 (Experimental): Subjects will be randomized to receive either GSK598809 25 mg or Placebo.
  Interventions: Drug: GSK598809; Drug: Placebo
- Subjects in Cohort-4 of Section 1 (Experimental): Subjects will be randomized to receive either GSK598809 40 mg or Placebo.
  Interventions: Drug: GSK598809; Drug: Placebo
- Subjects in Cohort-5 of Section 2 (Experimental): Subjects will be randomized to receive either ascending doses of GSK598809 75, 120 and 175 mg or Placebo. There will be a washout period of 6 days between the doses.
  Interventions: Drug: GSK598809; Drug: Placebo
- Subjects in Cohort-6 of Section 3 (Experimental): Subjects will receive caffeine on day -1 and after randomization subject will either receive GSK598809 or Placebo on Day 1. After washout period of 1-week subject will either receive GSK598809 or Placebo for 28 days.
  Interventions: Drug: GSK598809; Drug: Placebo; Drug: Caffeine

INTERVENTIONS:
Drug: GSK598809 — GSK598809 will be available as 5 and 25 mg capsules. Subjects will receive GSK598809 capsules orally with water.
  Other Names: GSK598809/Placebo
Drug: Placebo — Subjects will receive matching placebo capsules to GSK598809 orally with water.
Drug: Caffeine — Caffeine 100 mg will be available as oral solution or tablet and subjects will receive Caffeine 100 mg orally on -1 day. On Day 35 caffeine and GSK598809 will be co-administered.
  Arms: Subjects in Cohort-6 of Section 3

SUMMARY:
GSK598809 is being developed as an innovative treatment for substance dependence and potentially other compulsive behavioral disorders. This study will evaluate the safety, tolerability and pharmacokinetics of repeat doses of GSK598809 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female subject, aged 18-50 years inclusive.
* A female subject is eligible to participate if she is of Non-childbearing potential or Child-bearing potential and agrees to use adequate contraceptive methods until 90 days post-last dose.
* Body weight ≥50 kg and BMI within the range 18.5-29.9 kg/m2 inclusive.
* Healthy as judged by the responsible physician. No clinically significant abnormality in the medical, psychiatric or laboratory evaluation, including 12-lead ECG and 24-h Holter ECG.
* Signed and dated written informed consent before admission to the study.
* The subject is able to understand and comply with the Investigator's instructions and the requirements and restrictions of the protocol

Exclusion Criteria:

* The subject has a positive pre-study breath test for alcohol or smoking, or a positive urine drug screen. Drugs that will be screened for are amphetamines, barbiturates, cocaine, opiates, cannabinoids, benzodiazepines, PCP and cotinine.
* A positive result for Hepatitis B surface antigen, Hepatitis C antibody, or HIV 1/2 at the screening visit.
* Abuse of alcohol, defined as an average weekly intake of more than 28 units (males) or 21 units (females), or an average daily intake of more than 4 units. 1 unit is equivalent to half a pint (285 mL) of beer, 1 measure (25 mL) of spirits, or 1 glass (125 mL) of wine.
* Liver function tests (LFT) that are above the reference range at screening and that remain elevated when repeated (to be discussed with the sponsor, if necessary).
* Consumption of grapefruit juice or grapefruit within 7 days before the first dose of study medication and until collection of the final blood sample for pharmacokinetic analysis.
* Subject is not willing to eat the standard meals provided by the CPRU.
* Participation in other clinical trials of a new chemical entity or a prescription medicine, within the previous 3 months.
* Use of prescription or non-prescription medicines, including over-the-counter remedies, vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before the first dose of study medication, unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with the study procedures or compromise subject safety.
* Loss of more than 400 mL blood during the 3 months before the study, e.g. as a blood donor.
* History or presence of allergy to the study drug or drugs of this class, or a history of any other allergy that, in the opinion of the responsible physician, contraindicates the subject's participation.
* Regular use of tobacco- or nicotine-containing products within 6 months of the start of the study.
* Male subject does not agree to use a condom and spermicide during sexual intercourse with pregnant or lactating females; or if engaging in sexual intercourse with a female partner who could become pregnant. It is strongly recommended that in addition to this the female also uses another form of contraception. This criterion must be followed from the time of the first dose of study medication until 90 days after the last dose of study medication.
* History of a psychiatric diagnosis Axis I or Axis II (DSMIV), or presence of a current psychiatric diagnosis based upon psychiatric evaluation.
* History or presence of respiratory illnesses, gastrointestinal, hepatic or renal disease, or any condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Screening ECG with a QTc interval of >450 msec and/or a PR interval outside the range 120-220 msec inclusive, or an ECG that is not suitable for QT measurements
* Semi-supine vital signs at screening outside ranges defined in the protocol:
* Reduction, in systolic blood pressure, at screening, of 20 mm Hg or more on standing (compared with semi-supine measurement).
* Personal or family history of long QT syndrome or other cardiac conduction disorder, or other clinically significant cardiac disease.
* Serum electrolyte concentration outside the reference range.
* The subject has a serum prolactin that exceeds the normal range.
* Inability to abstain from strenuous physical activity for 24 h before screening, follow-up, and each admission to the ward.
* Presence or history of a recognised sleep disorder, or subject complains of sleep disturbances and/or is receiving treatment for sleep disorders, which might (on the basis of medical judgement) affect the pharmacodynamic or safety assessments.
* Inability to be successfully trained in tests of cognition. Additional Criteria for Section 3 only
* Consumption of coffee, cola or other caffeine containing drinks (Caffeine is one of the study substrates) within 4 days preceding the first dose
* Consumption of charcoal-broiled beef or cruciferous vegetables (e.g. broccoli, cabbage, brussel sprouts, cauliflower) within 7 days prior to the first dose . This foodstuff is a known inducer of the CYP1A2 enzyme

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2007-03-01 (Actual); Primary Completion 2008-08-22 (Actual); Study Completion 2008-08-22 (Actual)

PRIMARY OUTCOMES:
Safety measures: ECG, Vital Signs, Adverse Events for 48 hours after dosing. PK measures: Blood sampling for GSK598809 for upto 96hr post dose | Up to Day 39

SECONDARY OUTCOMES:
Tests on cognition (thinking) for 24 hours after dosing | Up to Day 36
Akathisia assessment | Up to Day 36
Involuntary Movements | Up to Day 36
Simpson Angus Scale (SAS) | Up to Day 36
Serum prolactin, GH and thyroid stimulating hormone (TSH), total and free testosterone, LH and FSH concentrations as possible | Up to Day 39
Psychological assessment | Up to Day 36
Cognition/impulsivity: | Up to Day 35
Pharmacokinetics: | Up to Day 38
GSK685249 levels to derive pharmacokinetic parameter | Up to Day 38

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- See also: Results for study DAN106587 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/DAN106587?search=study&search_terms=DAN106587#rs